CLINICAL TRIAL: NCT03468296
Title: Two-week Retreatment Interval Study for Treated Age-related Macular Degeneration Refractory to Monthly Aflibercept
Acronym: TRISTAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tennessee Retina (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-AMD-1819
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continued Q2 Week Treatment (Experimental): Will receive intravitreal aflibercept (2.0mg) injections for an additional four consecutive 2 week intervals at weeks 18, 20, 22, and 24
  Interventions: Drug: Intravitreal Aflibercept Injection 2mg
- Treat-And-Extend Treatment (Active Comparator): Will receive intravitreal aflibercept (2.0mg) injections on a treat-and-extend basis through week 24 with a minimum inter-treatment interval of q4 weeks.
  Interventions: Drug: Intravitreal Aflibercept Injection 2mg

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection 2mg — Aflibercept is a recombinant fusion protein consisting of portions of human VEGF receptors 1 and 2 extracellular domains fused to the Fc portion of human IgG1 formulated as an iso-osmotic solution for intravitreal administration.
  Other Names: Aflibercept; EYLEA®; VEGF Trap-Eye

SUMMARY:
This study is designed to evaluate the safety and efficacy of every 2 week intravitreal aflibercept injections in a population of neovascular AMD patients that have demonstrated refractory subretinal fluid with or without intraretinal fluid despite prior monthly intravitreal aflibercept treatment.

DETAILED DESCRIPTION:
Eligible patients will be scheduled to receive intravitreal aflibercept (2.0mg) injections for six consecutive 2 week (13-15 days) intervals with injections administered at weeks 0, 2, 4, 6, 8, 10, and 12. The primary endpoint visit to assess response to sustained q2week therapy will be at the week 14 visit. No treatment will be administered at this visit. All patients will then return at week 16 for the randomization visit and receive a repeat intravitreal aflibercept (2.0mg) injection. For purposes of randomization, patients will be separated into the following groups:

* Q2 week complete responders: absence of subretinal fluid on OCT at week 16
* Q2 week incomplete responders: persistent subretinal fluid on OCT at week 16

The "q2 week complete responders" will subsequently be transitioned to a treat and extend regimen with a minimum inter-treatment interval of 4 weeks through week 24. The "q2 week incomplete responders" will be randomized in a 1:1 fashion into one of two arms:

* Continued q2 week treatment: intravitreal aflibercept (2.0mg) injections for an additional four consecutive 2 week intervals at weeks 18, 20, 22, and 24
* Transition to treat-and-extend treatment: through week 24 with a minimum inter-treatment interval of q4 weeks. This arm is identical to regimen for "q2 week complete responders."

Beginning in week 24, all patients (all groups) will undergo treatment delivered on a treat-and-extend basis with a minimum inter-treatment interval of 4 weeks through the week 50. Patient visits will be treated no more frequent than q4 weeks during treat-and-extend portions of the protocol.

All patients will have a mandatory study termination visit at week 52 (-1/+2 weeks). No study treatment will be administered after week 50. Patients receiving a study treatment after week 48 will return 4 weeks after this final study treatment for study termination visit. Patients receiving a study treatment at or before week 48 in whom the treat-and-extend protocol would dictate a subsequent visit after week 52 will instead return at week 52 for a study termination visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* A diagnosis of choroidal neovascularization related to age-related macular degeneration
* ETDRS refracted BCVA ≥ 20/200
* Prior treatment with any anti-VEGF agent for ≥ 12 months
* Prior treatment with at least five intravitreal aflibercept at the time of screening (week -2) with an average inter-treatment interval <35 days
* Presence of persistent subretinal fluid with or without intraretinal fluid on OCT at most recent standard of care visit occurring 28-35 days following most recent intravitreal aflibercept injection
* Demonstration of definite improvement in overall retinal thickness and/or subretinal fluid on OCT based on evaluation of examining investigator at screening visit (week -2) 13-15 days following most recent standard of care visit

  o Note: screening OCT will be performed prior to dilation to allow for undilated ETDRS BCVA testing following confirmation of eligibility
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Ocular Exclusion Criteria:

* Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g. advanced diabetic retinopathy, advanced glaucoma)
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of macula-involving rhegmatogenous retinal detachment or macular hole (Stage 2 - 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia in the study eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)

Systemic Exclusion Criteria

* Use of systemic anti-VEGF medications within 6 months of screening visit
* History of cerebrovascular accident, myocardial infarction, ventricular arrhythmia, unstable angina, coronary or peripheral artery bypass or stenting within 6 months of day 0
* History of deep vein thrombosis or pulmonary embolus within 6 months of day 0
* Uncontrolled hypertension (>160/100 on medical treatment)
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception prior to the initial dose administration (baseline visit, week 0). Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

  * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through Week 14
  Frequency and severity of ocular and systemic adverse events

SECONDARY OUTCOMES:
Retinal Thickness | Weeks 14, 16, 24, 52
  Central Subfield Thickness on Optical Coherence Tomography
Subretinal Fluid Height | Weeks 14, 16, 24, 52
  Max subretinal fluid height week on Optical Coherence Tomography
Pigment Epithelial Detachment Height | Weeks 14, 16, 24, 52
  Max pigment epithelial detachment height on Optical Coherence Tomography
Proportion of Dry Maculas | Weeks 14, 16, 24, 52
  Proportion of eyes with a dry macula (no subretinal fluid on Optical Coherence Tomography)
Best-Corrected Visual Acuity | Weeks 14, 24, and 52
  Mean best-corrected visual acuity
Change in Best-Corrected Visual Acuity | Weeks 14, 24, and 52
  Mean change in best-corrected visual acuity from baseline
Proportion gaining >5 letters of Best-Corrected Visual Acuity | Weeks 14, 24, and 52
  Proportion of eyes gaining > 5 letters
Treatment Burden | Through Week 52
  Mean number of injections administered
Ability to Extend Treatment Interval | Through Week 52
  Proportion of eyes able to be extended during treat-and-extend dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Tennessee Retina, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider EW, Thomas MK, Recchia FM, Reichstein DA, Awh CC. SUSTAINED BIWEEKLY AFLIBERCEPT FOR REFRACTORY NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: The Prospective TRISTAR Study. Retina. 2023 May 1;43(5):739-746. doi: 10.1097/IAE.0000000000003729. PMID 36728874